CLINICAL TRIAL: NCT06942663
Title: Randomized Phase II Trial Evaluating DFS in the Absence of an Adjuvant Component of Perioperative Chemotherapy in Patients With Stage IB-III Gastric Cancer Who Achieved pCR or TRG4-5 on the Mandard Scale on Neoadjuvant Chemotherapy
Brief Title: Randomized Phase II Trial Evaluating DFS in The Absence of an Adjuvant Component of Perioperative Chemotherapy in Patients With Gastric Cancer
Acronym: JAGC1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nizhny Novgorod Regional Clinical Oncology Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JAGC - 1
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A ( patients with pCR - no adjuvant therapy ) (Experimental): Patients will not receive adjuvant chemotherapy
  Interventions: Other: Surveillance
- Group B ( patients with pCR - adjuvant therapy ) (Active Comparator): Patients will receive an adjuvant component of perioperative chemotherapy
  Interventions: Drug: Adjuvant Chemotherapy
- Group C ( patients with TRG of 4-5 - no adjuvant therapy ) (Experimental): Patients will not receive adjuvant chemotherapy.
  Interventions: Other: Surveillance
- Group D ( patients with TRG of 4-5 - adjuvant therapy ) (Active Comparator): Patients will receive an adjuvant component of perioperative chemotherapy
  Interventions: Drug: Adjuvant Chemotherapy

INTERVENTIONS:
Other: Surveillance — Close monitoring for disease recurrence.
  Arms: Group A ( patients with pCR - no adjuvant therapy ); Group C ( patients with TRG of 4-5 - no adjuvant therapy )
Drug: Adjuvant Chemotherapy — The adjuvant chemotherapy regimen will be standardized based on current clinical guidelines and may include combinations of agents such as fluoropyrimidines and oxaliplatin with or without docetaxel. Treatment until the progression of the process is detected or the maximum effect of therapy is achieved (the maximum duration of treatment is 3 months).
  Arms: Group B ( patients with pCR - adjuvant therapy ); Group D ( patients with TRG of 4-5 - adjuvant therapy )

SUMMARY:
This single-center, open-label, randomized phase II trial (JAGC-1) will evaluate whether adjuvant chemotherapy can be safely omitted in patients with stage IB-III gastric cancer (cT2-4a and/or N+) who have achieved a pathological complete response (pCR) or TRG 4-5 on the Mandard scale, following neoadjuvant chemotherapy and surgery. The study aims to compare disease-free survival and quality of life in patients receiving or not receiving adjuvant chemotherapy after neoadjuvant treatment and surgery.

DETAILED DESCRIPTION:
Population: patients with localized or locally advanced gastric cancer ( cT2-4a and/or N+ according to TNM, 8th revision, 2017) after having undergone the full extent of the planned neoadjuvant component of perioperative chemotherapy, radical surgical intervention, with a histological tumor regression grade classified as pCR or TRG 4-5 according to the Mandard scale

Study design Patients will be randomized in a ratio of approximately 1:1:

Patients who achieve pCR will be randomly assigned to one of two groups:

* Group A (no adjuvant therapy): Patients will not receive adjuvant chemotherapy
* Group B (adjuvant therapy): Patients will receive the adjuvant component of perioperative chemotherapy

Patients who achieve a TRG of 4-5 on the Mandard scale will be randomly assigned to one of two groups:

* Group C (adjuvant therapy): Patients will not receive adjuvant chemotherapy.
* Group D (no adjuvant therapy): Patients will receive the adjuvant component of perioperative chemotherapy.

Patients in the groups with adjuvant therapy will receive treatment until progression or maximal effect of therapy is detected (the longest duration of treatment is 3 months).

ELIGIBILITY:
Inclusion Criteria:

* - Obtaining informed consent to participate in the study.
* Morphologically confirmed gastric adenocarcinoma.
* The presence of localized or locally advanced gastric cancer (cT2-4a and/or N+)
* The full volume of the planned neoadjuvant component of perioperative chemotherapy was performed
* Radical surgical intervention was performed for the primary tumor of gastric cancer
* The histological degree of tumor regression after surgical resection was classified TRG1 and without metastasis to regional lymph nodes N0 or TRG 4-5 based on the Mandard tumor Regression scale.
* ECOG score 0 - I.
* Absence of severe uncontrolled concomitant chronic and acute diseases.
* Adequate liver and bone marrow function
* Neutrophils > 1.5*109/l
* Hemoglobin >85 g/l
* Platelets >100*109/l
* Increased transaminases and/or bilirubin < 2 art.

Exclusion Criteria:

* Lack of a neoadjuvant component of perioperative chemotherapy or insufficient number of courses
* The time after surgical treatment is more than 12 weeks
* Stage IV of the disease
* Her2-positive and/or MSI\dMMR stomach cancer
* Severe uncontrolled concomitant chronic or acute diseases
* The presence of a second malignant tumor (with the exception of previously cured malignant neoplasms)
* Any conditions that, in the opinion of the doctor, interfere with the examination procedures
* With incomplete tumor response to treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival rates | 3 years
  Comparison of 3-year DFS in the group receiving the adjuvant component of perioperative chemotherapy and in the group without it and comparison of the indicators of 3-year DFS with TRG 4-5 on the Mandard scale in the group receiving the adjuvant component of perioperative chemotherapy and in the group without it.

SECONDARY OUTCOMES:
Аssessment of the quality of life | 3 years
  Quality of life assessment by European Organisation for Research and Treatment of Cancer scale Quality of Life Questionnaire - Core 30 (QLQ-C30) by Scoring of the QLQ-C30 Summary Score using the descriptive analysis with the qlqc30 command (detailed description in manual ISBN 2-9300 64-22-6).

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Gamayunov, DMS, Study Director — RESEARCH INSTITUTE OF CLINICAL ONCOLOGY "NIZHNY NOVGOROD REGIONAL CLINICAL ONCOLOGICAL DISPENSARY"

IPD SHARING:
Plan to Share IPD: No